CLINICAL TRIAL: NCT05385861
Title: A Phase I/II Study of Nal-IRI (ONIVYDE® ) and Carboplatin in Patients With Advanced or Metastatic Gastroenteropancreatic Poorly Differentiated Neuroendocrine Carcinoma
Brief Title: Nal-IRI (ONIVYDE® ) and Carboplatin in Patients With Advanced or Metastatic GEP-NET
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); Chang Gung Memorial Hospital (Other); China Medical University Hospital (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2222
Record Dates: First submitted 2022-05-09; First posted 2022-05-23 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: GEP-NET
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor | interventions — irinotecan sucrosofate; Carboplatin

STUDY DESIGN:
Intervention Model Description: an investigator-initiated, single-arm phase 1/2 study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nal-IRI (ONIVYDE®) and Carboplatin (Experimental): nal-IRI (ONIVYDE®) and Carboplatin
  Interventions: Drug: nanoliposomal irinotecan plus carboplatin

INTERVENTIONS:
Drug: nanoliposomal irinotecan plus carboplatin — Dose in phase 1 cohort:
  Dose level 1= nanoliposomal irinotecan 100 mg/m2 plus carboplatin AUC=4, intravenously both on day 1, q3wk
  Dose level 0= nanoliposomal irinotecan 80 mg/m2 plus carboplatin AUC=4, intravenously both on day 1, q3wk
  Dose level -1= nanoliposomal irinotecan 60 mg/m2 plus carboplatin AUC=4, intravenously both on day 1, q3wk
  Carboplatin dose (mg) is calculated by the Calvert formula: AUC x (eGFR + 25). Cockcroft-Gault equation: eGFR (calculated Ccr)= [(140-age) x weight x 0.85 (if female)] / (72 x serum Cr). The maximum eGFR for dose calculation is 125 ml/min.
  In Phase 2 Cohort Patients will be treated until disease progression, unacceptable toxicity or other condition meeting the treatment discontinuation criteria.
  Other Names: Phase 1 cohort; Phase 2 Cohort

SUMMARY:
The current study is an investigator-initiated, single-arm phase 1/2 study that enrolled patients with advanced or recurrent and/or metastatic gastroenteropancreatic poorly differentiated neuroendocrine carcinoma for the treatment of nal-IRI (ONIVYDE®) plus carboplatin as the first-line chemotherapy.

DETAILED DESCRIPTION:
Eligible patients will be treated into two cohorts.

In adaptive phase 1 cohort:

Six patients will be enrolled in safety run-in cohort of dose level 0. If less than 2 patients experience dose-limiting toxicity (DLT) in dose level 0, dose level 1 will be tested. However, if more than 1 patients experience DLT in dose level 0, dose level -1 will be tested. The MTD at which no more than 1 of the 6 patients experience DLT will be determined for the phase 2 cohort. Otherwise, additional 6 patients will be tested in the dose level -1. Based on results from safety run-in cohort, PR2D will be determined. The evaluable patients in RP2D cohort will be incorporated into phase 2 cohort for final analysis.

Dose in phase 1 cohort:

Dose level 1= onivyde 100 mg/m2 plus carboplatin AUC=4, intravenously both on day 1, q3wk Dose level 0= onivyde 80 mg/m2 plus carboplatin AUC=4, intravenously both on day 1, q3wk Dose level -1= onivyde 60 mg/m2 plus carboplatin AUC=4, intravenously both on day 1, q3wk Carboplatin dose (mg) is calculated by the Calvert formula: AUC x (eGFR + 25). Cockcroft-Gault equation: eGFR (calculated Ccr)= [(140-age) x weight x 0.85 (if female)] / (72 x serum Cr). The maximum eGFR for dose calculation is 125 ml/min.

The definition of DLT:

Following toxicities occur during the first cycle of the combination chemotherapy with nal-IRI (ONIVYDE®) and carboplatin will be considered as DLTs. Toxicities are assessed by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).

* Grade 4 neutropenia (ANC < 500/μL) ≥3 days' duration under primary G-CSF support
* Grade 3 or higher neutropenia (ANC < 1,000/μL) with concurrent active infection requiring IV antibiotics treatment
* Grade 4 thrombocytopenia (platelet counts < 25,000/μL)
* Grade 3 thrombocytopenia (platelet counts < 50,000/μL) associated with active bleeding that transfusion is required
* Any grade 3 or higher treatment-related non-hematologic toxicity (except for anorexia/nausea, vomiting, and asthenia/fatigue)
* Any adverse drug reactions lead to more than 3 weeks delay

In Phase 2 Cohort Patients will be treated until disease progression, unacceptable toxicity or other condition meeting the treatment discontinuation criteria.

Tumor response will be assessed according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) every 6 weeks.

Adverse events (AEs) will be evaluated according to the National Cancer Institute's Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).

Patients sign additional consent to participate in the next generation sequencing study will be required to have extra tissue samplings at the study entry.

A follow-up visit is required approximately 30 days after treatment discontinuation. Overall survival status will be followed by clinic visit or by phone every 3 months until death or the maximum of 3 years, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed locally advanced or metastatic gastroenteropancreatic poorly differentiated neuroendocrine carcinoma.
2. patients either are chemotherapy-naive or had received adjuvant chemotherapy > 6 months before recurrence.
3. at least one measurable lesion according to the RECIST version 1.1..
4. patients were aged 20 to 80 years with ECOG performance status of 0 to 1.
5. patients had a life expectancy ≥ 3 months.
6. patients had adequate renal function with defined as serum creatinine ≤ 2 times the upper limit of normal (ULN) or eGFR (calculated Ccr) ≥ 45 mL/min.
7. patients had adequate hepatic function, defined as total bilirubin ≤ 1.5 times the ULN and alanine aminotransferase ≤ 2.5 the ULN and ≤ 5 times the ULN within the setting of liver metastases.
8. patients had adequate bone marrow function, defined as an absolute neutrophil count ≥ 1500/mm3, platelet count ≥ 100,000/mm3, and hemoglobin ≥ 9 g/dL.
9. Normal ECG or abnormal ECG without any clinical significantly findings.
10. Able to understand and sign an informed consent (or have a legal representative who is able to do so).

Exclusion Criteria:

1. a history of palliative chemotherapy or disease recurrence < 6 months from the time of last adjuvant chemotherapy and/or radiotherapy.
2. known hypersensitivity to liposome product, irinotecan or carboplatin.
3. receipt of major surgery within the past 4 weeks before study enrollment.
4. With clinically significant gastrointestinal disorder including bleeding, inflammation, occlusion or diarrhea > grade 2.
5. concurrent severe infection with intravenous systemic antibiotics treatment.
6. severe, uncontrolled medical condition including severe liver disease, heart disease, uncontrolled diabetes or hypertension, or pulmonary disease.
7. another previous malignancy diagnosed within the past 5 years except for nonmelanoma skin cancer or stage I cervical cancer.
8. active CNS metastasis defined by clinical symptoms, cerebral edema, steroid or anti-convulsant requirement, or progressive growth. Patients with a history of CNS metastasis or cord compression are allowed in the study if they have been treated and are clinically stable.
9. psychiatric illness or social situation that would preclude study compliance
10. women with pregnant or breast feeding (a urine pregnancy test must be performed on all patients who are of childbearing potential before entering the study, and the result must be negative).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
MTD and RP2D | 3 Years
  • in phase 1 cohort, to determine MTD (maximum tolerated dose) and recommended phase 2 dose (RP2D)
tumor response rate | 3 Years
  • in phase 2 cohort, to assess the objective tumor response rate

SECONDARY OUTCOMES:
PFS and OS | 3 Years
  • to assess other efficacy variables, including disease control rate, progression free survival (PFS), and overall survival (OS)
To explore the treatment-related adverse events as assessed by CTCAE v5.0 | 3 Years
  • Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-Wu Liu, Study Director — Taiwan Cooperative Oncology Group, NHRI
Locations (6):
- Taiwan (6):
  - Chang-Gung Memorial Hospital, Kaohsiung, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital (Lin-Kou),, Linkou District
  - China Medical University Hospital, Taichung
  - National Cheng-Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei